CLINICAL TRIAL: NCT03165487
Title: Differential Comparison of the Breast Tumor Microenvironment Between Luminal A and Triple Negative Breast Cancer With and Without Radiation Treatment
Brief Title: Comparison of the Breast Tumor Microenvironment
Status: Active, not recruiting | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Eileen Connolly, Assistant Professor, Columbia University
Other Study IDs: AAAO7708
Record Dates: First submitted 2017-05-22; First posted 2017-05-24 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Triple Negative Breast Cancer; Hormone Receptor Positive Malignant Neoplasm of Breast
Keywords: Triple Negative Breast Cancer; microenvironment; IORT; Hormone Receptor Positive, HER 2 negative
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Two specimens will be collected. A shaved margin of the area surrounding the tumor, considered as "normal" tissue, will be collected at two time points. The tissue will be collected prior to intraoperative radiation therapy, and immediately after. Blood will also be collected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Luminal A Breast Cancer: Luminal A Breast cancer subjects will have tissue specimens and blood collected before and after IORT during the Breast conserving surgery.
  Interventions: Other: Breast tissue collection; Other: Blood sample collection
- Triple Negative Breast Cancer: Triple Negative breast cancer subjects will have tissue specimens and blood collected before and after IORT during the Breast conserving surgery.
  Interventions: Other: Breast tissue collection; Other: Blood sample collection

INTERVENTIONS:
Other: Breast tissue collection — During Breast Conservation Surgery, one sample will be collected before and after IORT.
Other: Blood sample collection — Blood will be collected before and after IORT, and at the two week follow-up.

SUMMARY:
The goal of the project is to identify a molecular signature of tumor stroma from "normal" adjacent breast tissue obtained prospectively at the time of breast conserving surgery before and after receiving intraoperative radiation therapy (IORT) in subjects that have luminal A and triple negative breast cancer. IORT is considered as being standard of care.

DETAILED DESCRIPTION:
There is evidence that the normal tissue around a tumor plays a role in determining how the tumor behaves, including how it will respond to treatments and how likely it is to recur. In breast cancer, radiation is used to decrease the chance of recurrence in the area where the tumor is removed. This risk of recurrence varies between different types of breast cancer. The investigators seek to study the proteins produced in normal tissue surrounding breast tumors. The tissue will be taken from women who are receiving radiation to the breast at the time of their surgery (known as intraoperative radiation), one specimen taken before radiation and one after. A new process will be used to stabilize the tissue rapidly and allow the proteins to be identified before they break down. This will allow us to identify differences in the proteins produced by cells before and after radiation and between two types of breast cancers, luminal A (less likely to recur) and triple negative (more likely to recur). Identifying these differences in proteins may allow them to be used in the future as markers to predict the likelihood of tumors recurring.

ELIGIBILITY:
Inclusion Criteria:

* Female, age greater than or equal to 40
* Core biopsy proven invasive breast carcinoma or ductal carcinoma in situ (DCIS), all subtypes excluding invasive lobular carcinoma due to increased risk for multifocal disease
* Human epidermal growth factor receptor 2 (HER2) negative regardless of hormone receptor status
* Clinically less than or equal to 3cm unifocal lesion
* Clinically node negative
* Must have diagnostic mammogram performed within last 6 months
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) less than or equal to 1
* Appropriate renal, liver, and hematologic lab values
* Ability to give informed consent

Exclusion Criteria:

* Multifocal disease
* Clinically N1 disease at diagnosis
* Invasive lobular carcinoma
* Metastatic disease
* Patients for whom RT would be contraindicated (e.g., connective tissue disorder or prior ipsilateral breast radiation)
* Patients with known BRCA1/2 mutations
* Pregnant or nursing

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the outpatient Breast Surgery and Radiation Oncology Clinics of Columbia University
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with significant mean percent change in Tumor Infiltrating Lymphocytes (TILs) | Two weeks
  This outcome measure is designed to measure the amount of TILs in newly diagnosed luminal A and Triple Negative Breast Cancer (TNBC) tumors. The mean percent change in TILS in tumor tissue from initial core biopsy samples will be compared with pathology samples from definitive surgery after IORT between the two different breast cancer sub-types.

CONTACTS AND LOCATIONS:
Overall Officials: Eileen Connolly, MD, Principal Investigator — Assistant Professor of Radiation Oncology
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No